CLINICAL TRIAL: NCT06198166
Title: Effects of Cuevas Medek Exercises on Balance and Posture Control in Children With Autism Spectrum Disorder
Brief Title: Effects of Cuevas Medek Exercises Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/RCR&AHS/23/0752
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Balance; Cuevas Medek Exercises(CME)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Participants will get separate treatment protocol as and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuevas Medek (Experimental): This group will receive CME In a following procedure: supporting the patient in balance at the leg level and with slight posterior support. Then, once kept in the air for few seconds, slight up and down oscillations will make. These oscillations will reflexively induce an increase in tone of the body extensors, but also of the lower limbs. Always from the same position, gait movements will be imitated. At the beginning, due to poor coordination between muscle groups, the child may tend to go outside the support base and therefore we have to "run" following his center of gravity. The action is similar to the one when someone try to maintain balance of a cane in the palm and have to move his hands according to the cane's oscillation until he manage to regain balance
  Interventions: Other: Cuevas Medek
- Standard kinetic programs (Active Comparator): This group will receive standard kinetic programs consisting of stretching (2 sets 15 repetitions with 5 seconds hold) , passive mobilizations (2 sets of 20 repetitions), orthosis( for 6 hours). These techniques and orthotics devices typically focus on tight muscles, maintain proper foot alignment and to address sensory processing difficulties and promote relaxation. Stretching will focus on the hamstrings and calf muscles tightness.
  Interventions: Other: Standard kinetic programs

INTERVENTIONS:
Other: Cuevas Medek — Group A: will receive Cuevas Medek (CME) In a following procedure: supporting the patient in balance at the leg level and with slight posterior support. Then, once kept in the air for few seconds, slight up and down oscillations will make. The materials that will be used consists of three wooden boxes with the same dimensions (20cm x 40cm x 60cm), a bigger box, a wooden plate and two planks with the same dimensions (17cm x 80cm). Boxes
  Other Names: Standard
  Arms: Cuevas Medek
Other: Standard kinetic programs — Group B: will receive standard kinetic programs consisting of stretching (2 sets 15 repetitions with 5 seconds hold) , passive mobilizations (2 sets of 20 repetitions), orthosis( for 6 hours). These techniques and orthotics devices typically focus on tight muscles, maintain proper foot alignment and to address sensory processing difficulties and promote relaxation. Stretching will focus on the hamstrings and calf muscles tightness.
  Arms: Standard kinetic programs

SUMMARY:
Autism spectrum disorders (ASDs) describe a group of neurodevelopmental conditions in which the individuals face challenges with social engagement. This childhood disorder is characterized by core impairments in social/communication and repetitive behaviors. Autism spectrum disorder (ASD) is a lifelong disorder that occurs in approximately 1 in 68 children aged 8 years. It is primarily characterized by limited social interaction and communication, restricted interest, and stereotyped or repetitive behaviors. The motor deficits associated with ASD can relate to impairments of motor planning and control processes.

This Randomized Clinical Trial will recruit the participants through non probability convenience sampling. Participants will be randomly divided into 2 groups. Two groups of children aged between 2 and 6 years, suffering from autism spectrum disorder, one for control and one for experiment. Controlled will get conventional treatment while study group will get conventional treatment with Cuevas Medak Exercises (CME). Treatment duration is of 12 weeks. Progress will be monitored every month. The frequency of recovery sessions will 3 sessions/week, and the duration of a session will 45 minutes. Patient evaluation will be made at the beginning and the end of the treatment through pediatric balance scale and posture and postural ability scale. Data will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) describe a group of neurodevelopmental conditions in which the individuals face challenges with social engagement. This childhood disorder is characterized by core impairments in social/communication and repetitive behaviours. Two groups of children aged between 2 and 6 years, suffering from autism spectrum disorder, one for control and one for experiment. Controlled will get conventional treatment while study group will get conventional treatment with Cuevas Medak Exercises (CME). Treatment duration is of 12 weeks. Progress will be monitored every month. The frequency of recovery sessions will 3 sessions/week, and the duration of a session will 45 minutes. Patient evaluation will be made at the beginning and the end of the treatment through pediatric balance scale and posture and postural ability scale. Data will be analyzed through SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Children with medical diagnosis of mild ASD diagnosed by CARS assessment tool with score ranges from 15 to 30.
* Children having postural and balance problems with scoring of 8 out of 14 items of pediatric balance scale.
* Age ranging from 2 to 6 years
* Parental/Caregiver report of Difficulty with motor planning, motor skills and/or postural control.
* Children who will able to follow verbal instruction and participate in exercise program.

Exclusion Criteria:

* Children with planned surgical or medical surgeries during study period.
* Severe behavioral problems.
* Unstable medical condition.
* History neurological disorder (seizures, epilepsy)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | 12 weeks
  This tool is used for assessing change from baseline. The PBS is easy to administer, does not require specialized equipment, and can be completed in <20 minutes. A 0 to 4 grading scale provides a quantitative and qualitative measure of performance. It involves 14 mobility tasks, with the tasks varying in degrees of difficulty. The tasks are divided in to 3 domains, sitting balance, standing balance and dynamic balance. The PBS has high validity and reliability of 0.98. 41-56=low fall risk, 21-40 = medium fall risk, 0-20 high fall risk.
Posture and posture ability scale | 12 weeks
  The Posture and Postural Ability Scale is a 7-point ordinal scale for the assessment of postural ability in standing, sitting, supine and prone. There are six items for assessment of quality of posture in the frontal plane and another six items in the sagittal plane. The Cronbach alpha value of posture and postural ability scale is 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Intsam Aslam, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memari AH, Panahi N, Ranjbar E, Moshayedi P, Shafiei M, Kordi R, Ziaee V. Children with Autism Spectrum Disorder and Patterns of Participation in Daily Physical and Play Activities. Neurol Res Int. 2015;2015:531906. doi: 10.1155/2015/531906. Epub 2015 Jun 15. PMID 26171247